CLINICAL TRIAL: NCT01406925
Title: A Randomised, Placebo-controlled, Double-blind, Cross-over Study in Healthy Men and Women to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Intra-anal Doses of NRL001 for Three Doses Using a Cream Formulation Relative to a Matched Placebo Formulation for Reference
Brief Title: Safety and Tolerability of a Single Intra-anal Dose of NRL001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Hans-Jurgen Gruss, Norgine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRL001-02/2006(SD)
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo control
- Low dose NRL001 (Experimental): 0.5% NRL001 cream
  Interventions: Drug: NRL001 cream
- Intermediate dose NRL001 (Experimental): 0.75% NRL001 cream
  Interventions: Drug: NRL001 cream
- High dose NRL001 (Experimental): 1.0% NRL001 cream
  Interventions: Drug: NRL001 cream

INTERVENTIONS:
Drug: Placebo control — Placebo cream
  Arms: Control
Drug: NRL001 cream — Cream for single-dose intra-anal application
  Arms: High dose NRL001; Intermediate dose NRL001; Low dose NRL001

SUMMARY:
This study is conducted to explore the safety and tolerability and plasma pharmacokinetics of NRL001 after single intra-anal dose of 1mL cream at increasing concentrations.

ELIGIBILITY:
Inclusion Criteria:

IN.1) sex: male and female (non-child-bearing potential or using medically adequate contraception

IN.2) race: Caucasian

IN.3) BW: 50 - 100 kg

IN.4) BMI: 20 - 28 kg.m-2

IN.5) age: 21 - 50 years

IN.6) type: healthy on the basis of specified criteria evaluated at the screening visit

IN.7) willing and able to provide informed consent

Exclusion Criteria:

General

EX.1) Previous participation in the trial

EX.2) Participant in any other trial during the last 90 days

EX.3) Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months

EX.4) History of any clinically relevant allergy (including hypersensitivity to the trial medications)

EX.5) Presence of acute or chronic infection

EX.6) Presence or history of any relevant co-morbidity

EX.7) Resting systolic blood pressure > 140 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg

EX.8) Clinically relevant ECG-abnormalities, prolonged QTc with > 450 msec in males and > 460 msec in females in particular

EX.9) Presence of any relevant abnormality in the laboratory safety tests, especially low haemoglobin, increased liver enzymes

EX.10) Positive serology for HBsAg, anti HBc and anti HCV

EX.11) Positive HIV test

EX.12) Positive alcohol or urine drug test on recruitment (and upon admission)

EX.13) History of alcohol and/or drug abuse and/or daily use of > 30 gr alcohol

EX.14) Smoking more than 15 cigarettes/day or equivalent of other tobacco products

EX.15) Use of prohibited medication

EX.16) Suspicion or evidence that the subject is not trustworthy and reliable

EX.17) Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard

General - all females

EX.18) Positive pregnancy test

EX.19) Lactating

EX.20) Not using appropriate contraception in pre-menopausal women (note: under the conditions of the present study, women using hormonal contraceptives will be informed that this method is not sufficient during the study and that further i.e. mechanical methods [condom, diaphragm with spermicidal gel] should be used in addition).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Cmax of NRL001 | 30 mins, 1, 2, 3, 4, 5, 6, 8 and 12 hours after dosing

SECONDARY OUTCOMES:
AUC of NRL001 | 30 mins, 1, 2, 3, 4, 5, 6, 8 and 12 hours after dosing
Tolerability of NRL001 | Up to 12 hours post-dosing
  Spontaneously reported adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gruss, MD PhD, Study Director — Norgine
Locations (1):
- University Hospital MHAPT Zaritza Johanna, Sofia, Bulgaria